CLINICAL TRIAL: NCT05208944
Title: A Multicenter, Open-Label, Dose-Finding, Phase 2 Study Evaluating THIO Sequenced With Cemiplimab (LIBTAYO®) in Subjects With Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: THIO Sequenced With Cemiplimab in Advanced NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Maia Biotechnology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: THIO-101; 2023-504595-26-00 (EU CTIS Number); 2021-005136-34 (EudraCT Number)
Record Dates: First submitted 2021-12-05; First posted 2022-01-26 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: SQUAMOUS CELL CARCINOMA; ADENOCARCINOMA; LARGE CELL CARCINOMA; Carcinoma, Non Small Cell Lung; Carcinomas, Non-Small-Cell Lung; Lung Carcinoma, Non-Small-Cell; Lung Carcinomas, Non-Small-Cell; Non-Small-Cell Lung Carcinomas; Non-Small-Cell Lung Carcinoma; Carcinoma, Non-Small Cell Lung; Non-Small Cell Lung Carcinoma; Non-Small Cell Lung Cancer; Nonsmall Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Squamous Cell; Adenocarcinoma; Carcinoma, Large Cell | interventions — alpha-2'-deoxythioguanosine; cemiplimab

STUDY DESIGN:
Intervention Model Description: * Part A (Completed enrolment, N=10): Modified 3+3 design safety lead-in study of THIO 360 mg per cycle (120 mg on Days 1-3, sequenced with cemiplimab).
  * Part B (Completed enrolment, N=69): Randomized, dose-finding, Simon's 2-stage design, 3-arm study (THIO 60 mg, THIO 180 mg, or THIO 360 mg per cycle; all dose levels sequenced with cemiplimab), with optional extension cohort(s).
  * Revised Part C (Planned; N-37-48): all enrolled subjects will receive THIO 60 mg administered by 30-minute IV infusions once daily on Days 1-3 of every 3-week cycle (for a total of 180 mg per cycle). In addition, subjects randomized to the sequential combination arm (Arm 1), and subjects enrolled into the Arm 1 Expansion Cohort will also receive a fixed dose of cemiplimab (350 mg IV) on Day 5 of each
  * Part D (Planned; N=100): Single-arm Efficacy cohort evaluating the efficacy and safety of THIO 180 mg per cycle sequenced with cemiplimab as third-line treatment in patients with advanced/metastatic NSCLC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part A (Experimental): Safety lead-in, modified 3+3 design. Part A:
  Cohort 1: THIO total 360 mg per cycle (120 mg on Days 1-3 Q3W) plus 350 mg cemiplimab on Day 5; Cohort 2 (pending emerging data from Cohort 1): THIO total 180 mg per cycle (60 mg on Days 1-3 Q3W) plus 350 mg cemiplimab on Day 5
  Interventions: Drug: 6-Thio-2'-Deoxyguanosine; Drug: Cemiplimab
- Part B (Experimental): Cohort 1: THIO total 60 mg per cycle (20 mg on D1-3 Q3W) plus 350 mg cemiplimab on Day 5; Cohort 2: THIO total 180 mg per cycle (60 mg on D1-3 Q3W) plus 350 mg cemiplimab on Day 5; Cohort 3 (pending emerging data from Part A): THIO total 360 mg per cycle (120 mg on Days 1-3 Q3W) plus 350 mg cemiplimab on Day 5
  Interventions: Drug: 6-Thio-2'-Deoxyguanosine; Drug: Cemiplimab
- Part C (Experimental): To obtain clinical evidence of the efficacy and safety of the sequential combination of THIO 180 mg per cycle plus cemiplimab compared to single-agent THIO 180 mg per cycle as third-line treatment in subjects with advanced/metastatic NSCLC.
  Interventions: Drug: 6-Thio-2'-Deoxyguanosine; Drug: Cemiplimab
- Part D (Experimental): To determine the efficacy of THIO 180 mg per cycle (60 mg on Days 1-3, sequenced with cemiplimab) when administered as third-line treatment in subjects with advanced/metastatic NSCLC.
  Interventions: Drug: 6-Thio-2'-Deoxyguanosine; Drug: Cemiplimab

INTERVENTIONS:
Drug: 6-Thio-2'-Deoxyguanosine — small molecule telomere targeting agent
  Other Names: 6-thio-dG; THIO
Drug: Cemiplimab — programmed cell death protein 1 (PD-1) inhibitor
  Other Names: LIBTAYO®

SUMMARY:
THIO is a first-in-class small molecule telomere targeting agent, in development for the treatment of non-small cell lung cancer (NSCLC) in combination with cemiplimab (LIBTAYO®). THIO is preferentially incorporated into telomeres sequence in telomerase-positive cells leading to rapid telomere uncapping, genomic instability, and cell death.

Cemiplimab is a programmed cell death protein 1 (PD-1) inhibitor recently approved as a first-line treatment for patients with locally advanced or metastatic NSCLC with 50% or more PD-L1 expression. It is hypothesized that THIO administration prior to cemiplimab would restore tumor responses to immunotherapy in subjects who either developed resistance or relapsed after receiving first line treatment with an immune check point inhibitor.

DETAILED DESCRIPTION:
The THIO-101 study evaluates the safety and efficacy of different doses of THIO sequenced with fixed dose of cemiplimab (referred to as investigational products [IP]) in subjects with advanced NSCLC who progressed, discontinued due to toxicity, or relapsed after receiving prior therapy with an anti-PD-1/PD-L1 agent.

This study is a Phase 2, open-label, multicenter study comprised of 4 parts:

* Part A (Completed enrolment, N=10): Modified 3+3 design safety lead-in study of THIO 360 mg per cycle (120 mg on Days 1-3, sequenced with cemiplimab).
* Part B (Completed enrolment, N=69): Randomized, dose-finding, Simon's 2-stage design, 3-arm study (THIO 60 mg, THIO 180 mg, or THIO 360 mg per cycle; all dose levels sequenced with cemiplimab), with optional extension cohort(s).
* Revised Part C (Planned; N= 37 to 48)
* Part D (Planned; N=100): Single-arm Efficacy cohort evaluating the efficacy and safety of THIO 180 mg per cycle sequenced with cemiplimab as third-line treatment in patients with advanced/metastatic NSCLC.

This study aims to establish THIO followed by cemiplimab as a potential treatment regimen in a high unmet medical need setting.

A Safety Review Committee (SRC) will monitor subject safety during the study and will make recommendations to the Sponsor regarding enrollment, eg, de-escalating dose in Part A, proceeding to Part B, expanding an arm in Part B, opening Part C, and Part D of the study based on emerging data from prior study parts.

In each study part, on Cycle 1, Day 1, eligible subjects initiate treatment with THIO (at doses described for each study part below) as intravenous (IV) infusion, once daily, on Days 1-3 of every 3-week cycle (Q3W) followed by a fixed dose of cemiplimab (350 mg IV) on Day 5 Q3W. The only exception is the randomized Arm 2 of Part C, where subjects will be receiving single agent THIO (without sequential cemiplimab). Study treatment may continue until PD, occurrence of an unacceptable toxicity, withdrawal of consent, death, or two years on treatment, whichever occurs first.

The initial radiographic imaging for baseline assessment is to be conducted by the investigator up to 28 days before the first dose of THIO for tumor evaluation and measurements. The on-treatment radiographic assessments are to be performed every 2 cycles (every 6 weeks, ± 7 days) during the first year of treatment, and then every 3 cycles (every 9 weeks, ± 14 days) during the second year of treatment until documented PD, initiation of a new anti-cancer treatment, or completion of follow-up, whichever occurs first. The radiographic scans are to be assessed by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and/or iRECIST until PD, initiation of a new anti-cancer treatment, or end of the study, whichever occurs first. In Part D of the study, radiographic scans will also be assessed by a blinded independent central review (BICR) committee. Confirmation of CR and PR per RECIST v1.1 by consecutive radiographic imaging (computed tomography [CT]/magnetic resonance imaging [MRI]; same modality to be used for a given subject throughout the study) assessment 4-8 weeks from the date of first documentation is required. In Parts A, B, and C, radiographic scans are/will be collected and held for possible future retrospective independent evaluation.

To account for tumor pseudoprogression or delayed response with anti-PD1/PD-L1 immunotherapies, subjects may continue to receive IP beyond RECIST v1.1 defined progression at the discretion of the investigator and be assessed at a subsequent tumor assessment time point (≥ 4 weeks after the date of initial documentation of disease progression) to confirm PD according to iRECIST. Subjects must be consented to receive the IP beyond the initial progression and will discontinue IP once the progression is confirmed by iRECIST.

Safety assessments for all study patients (Parts A, B, C, and D) during each treatment cycle include complete or abbreviated physical examinations, routine safety laboratory testing (hematology, clinical chemistry, coagulation), thyroid hormone testing, vital sign evaluations, and electrocardiograms (ECGs).

All subjects will undergo end of treatment (EoT) visit 30 days post last treatment with IP. Subjects will be followed every 3 months until death, withdrawal of consent, loss to follow-up, or study termination by the Sponsor, whichever occurs first. Long-term follow-up can be via clinic visit, phone call to the subject or referring physician, or other method deemed appropriate by the site and should assess survival, progression, subsequent anti-cancer therapy and response. Any subject who discontinues treatment for reasons other than disease progression will continue to have radiographic assessments per standard of care and no less than every 3 months for the first year, and then every 6 months until documented disease progression, initiation of a new anti-cancer treatment, or end of follow-up. Subjects in Parts A and B only who discontinued treatment due to disease progression per RECIST 1.1 and did not receive post-progression treatment could be asked to complete standard of care radiographic assessments every 3 months for up to 1 year and then every 6 months until initiation of a new anti-cancer treatment or completion of follow-up. Response assessment in follow-up will include at minimum the modality used to determine response.

ELIGIBILITY:
Inclusion Criteria Age

1. At least 18 years of age at the time of signing the Informed Consent Form (ICF) prior to initiation of any study specific activities/procedures.

   Type of Subject and Disease Characteristics
2. Stage 3 or 4 histologically or cytologically confirmed NSCLC which has progressed or relapsed after treatment in the advanced setting

   ○ Stage 4 subjects: Part A and Part B: must have progressed or relapsed after first line treatment. Part C and Part D: must have progressed, discontinued due to toxicity, or relapsed after receiving (only) two prior lines of treatment for NSCLC in the advanced setting.

   ○ Stage 3 subjects - must have already failed, or be ineligible for, local, curative-intent therapy including surgery, and/or chemoradiation. Stage 3 subjects with documented relapse/progression after consolidation therapy with durvalumab following definitive chemoradiotherapy are eligible.
3. Subjects must have secondary resistance to the prior ICI, as defined by the Society for Immunotherapy of Cancer (SITC) Immunotherapy Resistance Task Force (IRTF) (Kluger 2020):

   Resistance phenotype Drug exposure requirements Best response Confirmation scan for PD requirement Confirmation scan timeframe Secondary resistance ≥ 6 months CR, PR, SD for > 6 months Yes [1] At least 4 weeks after disease progression (per RECIST V1.1) Other than when tumor growth is very rapid, and subjects are deteriorating clinically.

   Abbreviations: CR=complete response; PD=progressive disease; PR=partial response; SD=stable disease Note: Subjects with drug exposure > 6 weeks who achieved a PR or CR then progressed before 6 months, would still be eligible.
4. Part A and Part B: Only one prior treatment for NSCLC in the advanced setting, which must have included one anti-PD-1/PD-L1 agent with documented radiographic disease progression on or after treatment.

   * Prior treatment may have been with anti-PD-1/PD-L1 agent either alone or in combination with a non-anti-PD-1/PD-L1 treatment (e.g., chemotherapy)
   * Prior platinum-based chemotherapy is not required for eligibility.
   * Subjects receiving more than one ICI in the advanced setting (e.g., anti-PD-1/PD-L1 and anti-CTLA-4 compounds) will not be eligible.

   Part C and Part D: Only two prior treatments for NSCLC in the advanced setting, which must have included an anti-PD-1/PD-L1 agent, a platinum-based chemotherapy, and docetaxel, regardless of order or combination, with documented radiographic disease progression, intolerable toxicity, or relapse after treatment.

   ○ Combination of immune therapy is allowed (e.g., anti-PD-1/PD-L1 and anti-CTLA-4 compounds; anti-PD-1/PD-L1 and T-cell immunoreceptor with immunoglobulin and immunoreceptor tyrosine-based inhibition motif domain (TIGIT)-based immunotherapy).
5. No prior targeted therapy for driver mutations.
6. At least one measurable target lesion that meets the definition of RECIST v1.1.
7. Part A and Part B: An archival tissue sample (formalin fixed paraffin-embedded [FFPE] tissue block or unstained slides) is required if tissue is available at baseline. Sample does not need to be received by central lab prior to Cycle 1, Day 1 (C1D1). Subjects without archival tissue available at baseline may be eligible with Medical Monitor approval.

   Part C and Part D: Archival tissue is not required. Diagnostic Assessments
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
9. Demonstrate adequate organ function as defined below. All screening laboratories should be performed up to 14 days before initiating IP:

   Bone marrow function:

   ○ Neutrophil count ≥ 1500/mm3, hemoglobin ≥ 9.0 g/dL, platelet count ≥ 100,000/mm3

   Liver function:
   * Total bilirubin ≤ 1.5 x the upper limit of normal (ULN), up to ≤ 3 × ULN due to Gilbert's syndrome
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 1.5 × ULN. For subjects with liver metastases present at baseline, ALT and/or AST ≤ 3 × ULN is permitted.

   Renal function:

   ○ Creatinine clearance ≥ 60 mL/min calculated by the Cockcroft-Gault formula using actual body weight (see Table 15) or 24-hour urine collection.

   Gender and Reproductive Considerations
10. Women of childbearing potential (WOCBP) must have negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 72 hours prior to receiving the first administration of IP.
11. Contraception use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. Refer to Appendix 4, Section 10.4 for details and definitions of WOCBP, postmenopausal females and contraception guidance.
12. WOCBP must agree to use a highly effective birth control and refrain from oocyte donation during the study (prior to the first dose with THIO, for the duration of the treatment with THIO plus 6 months after last dose of IP), if conception is possible during this interval.
13. Male subjects and WOCBP partners of male subjects should use a combination of the methods specified in Section 10.4 for the women along with a male condom from first dose of THIO (Cycle 1, Day 1), for the duration of the treatment with THIO plus 6 months after last dose of IP, unless permanently sterile by bilateral orchidectomy. Male subjects should also refrain from sperm donation during this time.

    Informed Consent
14. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and in this protocol

Exclusion Criteria

1. Have not recovered from adverse events (must be Grade ≤ 1) due to prior anti-cancer treatment.
2. Untreated or symptomatic central nervous system (CNS) metastases. Note: subjects with treated asymptomatic brain metastasis are eligible.
3. Active gastrointestinal bleeding as evidenced by either hematemesis or melena.
4. History of another concurrent malignancy other than the present condition (except nonmelanoma skin cancer or carcinoma in situ of the cervix), unless in complete remission and off all therapy for that disease for a minimum of 3 years.
5. A condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids, adrenal replacement doses 10 mg daily prednisone equivalents, and systemic corticosteroids to manage adverse events (AEs) are permitted in the absence of active autoimmune disease.
6. Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy within 2 weeks of screening.
7. Positive for Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies), active hepatitis B or hepatitis C.
8. Significant cardiovascular impairment (history of New York Heart Association Functional Classification System Class III or IV) or a history of myocardial infarction or unstable angina within the past 6 months prior to IP initiation.

   a) QTcF > 480 msec at screening (based on average of triplicate ECGs at baseline).

   i. If the QTc is prolonged in a subject with a pacemaker or bundle branch block, the subject may be enrolled in the study if confirmed by the Medical Monitor.
9. Ongoing immune-related/stimulated adverse events (irAEs) from other agents or required permanent discontinuation of prior ICIs due to irAEs. Subjects with resolved irAE may be allowed to enroll following consultation with Sponsor's Medical Monitor (or designee).
10. Active autoimmune diseases or history of autoimmune diseases that may relapse, with the following exceptions:

    * Controlled type 1 diabetes;
    * Hypothyroidism (provided it is managed with hormone replacement therapy only);
    * Controlled celiac disease;
    * Skin diseases not requiring systemic treatment (e.g., vitiligo, psoriasis, or alopecia);
    * Any other disease that is not expected to recur in the absence of external triggering factors.
11. Pregnancy or lactating.
12. A serious nonmalignant disease (e.g., psychiatric, substance abuse, uncontrolled intercurrent illness, etc.) that could compromise protocol objectives in the opinion of the investigator and/or the Sponsor.
13. Any other condition that, in the opinion of the investigator, would prohibit the subject from participating in the study.

    Prior Therapy
14. Part C and Part D: more than two prior systemic treatments for advanced disease.
15. Prior chemotherapy and/or non-biologic targeted therapy within 4 weeks, or biologic targeted therapy, immunotherapy, and/or radiation therapy within 6 weeks prior to Cycle 1 Day 1. Subjects who receive targeted radiation therapy for localized palliative care may be eligible to start treatment < 6 weeks with Medical Monitor agreement.
16. Part A and Part B: Prior treatment with cemiplimab. Note: Part C and Part D: prior cemiplimab is permitted.
17. For subjects who have received prior treatment with an ICI: primary resistance to prior ICI therapy, as defined by the SITC IRTF (Kluger 2020):

    Resistance phenotype Drug exposure requirements Best response Confirmation scan for PD requirement Confirmation scan timeframe Primary resistance ≥ 6 weeks PD; SD for < 6 months Yes [1] At least 4 weeks after initial disease progression (per RECIST v1.1) [1] Other than when tumor growth is very rapid, and subjects are deteriorating clinically.

    Abbreviations: CR=complete response; PD=progressive disease; PR=partial response; SD=stable disease Note: Subjects with drug exposure > 6 weeks who achieved a partial or complete response then progressed before six months, would still be eligible.
18. Undergone major surgery within 4 weeks prior to Cycle 1, Day 1.
19. Received blood, red blood cell or platelet transfusion within 2 weeks before the first dose of IP.
20. Any live, attenuated, inactivated or research vaccines within 30 days prior to the first dose of IP. Refer to Section 6.9.1 for prohibited vaccines. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed.
21. Prior allogeneic hematopoietic stem cell transplant or solid organ transplant. Prior/Concurrent Clinical Study Experience
22. Currently enrolled in a clinical study involving another IP or nonapproved use of a drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.

    Other
23. History of allergy to excipients of THIO or cemiplimab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Estimated)
Dates: Start 2022-06-08 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To determine the safety and tolerability of THIO administered in sequence with cemiplimab in subjects with advanced NSCLC | Up to 2 years
  Part A: Incidence of DLTs
To assess the efficacy of THIO administered in sequence with cemiplimab in subjects with advanced NSCLC | Up to 2 years
  ORR, defined as the proportion of subjects with either a CR or PR, as assessed by the investigator based on RECIST v1.1
To assess the efficacy of THIO administered in sequence with cemiplimab in subjects with advanced NSCLC | Up to 2 years
  DCR defined as the proportion of subjects with CR, PR, or SD, as assessed by the investigator based on RECIST v1.1
To determine the safety and tolerability of THIO administered in sequence with cemiplimab in subjects with advanced NSCLC | Up to 2 years
  Part A: Incidence of DLTs Part A and Part B: Incidence of SAEs overall, by severity, by relationship to THIO and/or cemiplimab, and those that led to discontinuation of THIO and cemiplimab and/or withdrawal from study
To determine the safety and tolerability of THIO administered in sequence with cemiplimab in subjects with advanced NSCLC | Up to 2 years
  Part A and Part B: Incidence of TEAEs overall, by severity, by relationship to THIO and/or cemiplimab, and those that led to discontinuation of THIO and cemiplimab and/or withdrawal from study

SECONDARY OUTCOMES:
Additional efficacy evaluation | Up to 2 years
  Parts A, B, C and D: Duration of Response (DoR)
Safety Parts C and D To determine the safety and tolerability of THIO administered in sequence with cemiplimab in subjects with advanced/metastatic NSCLC | Up to 2 years
  Incidence of TEAEs (overall, by severity, by relationship to THIO and/or cemiplimab).
Additional efficacy evaluation | Up to 2 years
  Parts A, B, C and D: Progression Free Survival (PFS)
Additional efficacy evaluation | Up to 2 years
  Parts A, B, C and D: Overall Survival (OS)
Additional efficacy evaluation | Up to 2 years
  Parts C and D: Disease Control Rate (DCR) as assessed by the investigator based on RECIST 1.1
Additional efficacy evaluation | Up to 2 years
  Parts A, B, and C: Objective Radiographic Response Rate (ORR) defined as the proportion of subjects with either a CR or PR, as assessed by the investigator based on RECIST v1.1
Additional efficacy evaluation | Up to 2 years
  Part D: Objective Radiographic Response Rate (ORR) defined as the proportion of subjects with a confirmed CR or PR, as assessed by BICR based on RECIST v1.1.
Safety Parts C and D To determine the safety and tolerability of THIO administered in sequence with cemiplimab in subjects with advanced/metastatic NSCLC | Up to 2 years
  Incidence of treatment-emergent SAEs.
Safety Parts C and D To determine the safety and tolerability of THIO administered in sequence with cemiplimab in subjects with advanced/metastatic NSCLC | Up to 2 years
  Incidence of TEAEs of special interest
Safety Parts C and D To determine the safety and tolerability of THIO administered in sequence with cemiplimab in subjects with advanced/metastatic NSCLC | Up to 2 years
  Incidence of TEAEs leading to dose modifications or discontinuation of treatment.
Safety Parts C and D To determine the safety and tolerability of THIO administered in sequence with cemiplimab in subjects with advanced/metastatic NSCLC | Up to 2 years
  Incidence of and fatal TEAEs.

OTHER OUTCOMES:
To determine the PK of THIO and assess THIO PK / pharmacodynamics (PDy) exposure-response relationship | Up to 2 Years
  THIO concentration levels and PK parameters
Investigator-assessed anti-tumor activity of THIO sequenced with cemiplimab based on iRECIST | Up to 2 Years
  iORR as assessed by the investigator based on iRECIST
To assess blood biomarkers | Up to 2 years
  Blood level of interleukin (IL-6)
To evaluate anti-tumor activity of THIO and cemiplimab by the Investigator based on modified RECIST v1.1 for immune-based therapeutics (iRECIST) | Up to 2 years
  iRECIST Disease Control Rate (iDCR)
To assess PDy Parameters | Up to 2 years
  Gamma-H2AX in circulating tumor cells (CTCs) in blood
To assess PD7 Parameters | Up to 2 years
  PD-L1 levels in circulating tumor cells (CTCs) in blood
To assess blood biomarkers | Up to 2 years
  Blood level of c-reactive protein (CRP)
To assess blood biomarkers | Up to 2 years
  Blood level of CEA
To evaluate anti-tumor activity of THIO and cemiplimab by the Investigator based on modified RECIST v1.1 for immune-based therapeutics (iRECIST) | Up to 2 years
  iRECIST Objective Radiographic Response (iORR)
To evaluate anti-tumor activity of THIO and cemiplimab by the Investigator based on modified RECIST v1.1 for immune-based therapeutics (iRECIST) | Up to 2 years
  iRECIST Progressive Free Survival (iPFS)
To evaluate anti-tumor activity of THIO and cemiplimab by the Investigator based on modified RECIST v1.1 for immune-based therapeutics (iRECIST) | Up to 2 years
  iRECSIT Duration of Response iDoR

CONTACTS AND LOCATIONS:
Overall Officials: Victor Zaporojan, MD, Study Chair — Maia Biotechnology
Locations (33):
- Australia (3):
  - Sunshine Coast Haematology and Oncology Clinic, Buderim, Queensland
  - Cancer Research SA, Adelaide, South Australia
  - St. Vincent Hospital Melbourne, Fitzroy, Victoria
- Bulgaria (4):
  - MHAT "HEART AND BRAIN" EAD Clinic of Medical Oncology, Pleven
  - MC Synexus Sofia EOOD, Sofia
  - MHAT "Serdika" EOOD, Sofia
  - UMHAT "Sofiamed", Sofia
- Hungary (8):
  - Semmelweis Egyetem Pulmonologiai Klinika, Budapest
  - Országos Korányi Pulmonológiai Intézet, Budapest
  - Orszagos Onkologiai Intezet, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Tudogyogyaszati Klinika, Debrecen
  - Bács-Kiskun Megyei Oktatókórház, Onkoradiológiai Központ, Kecskemét
  - Mátrai Gyógyintézet, Mátraháza
  - Hetenyi Geza Korhaz, Onkologiai Kozpont, Szolnok
  - Tüdőgyógyintézet Törökbálint, Onkológiai Osztályc, Törökbálint
- Poland (9):
  - NZOZ FORMED 2 Sp. z o.o., Oświęcim, Oswiecim
  - Centrum Onkologii im. prof. F. Lukaszczyka, Bydgoszcz
  - Krakowski Szpital Specjalistyczny im. Jana Pawla II Oddzial Onkologii z Pododdzialem Diagnostyki Nowotworow Klatki Piersiowej, Krakow
  - Centrum Terapii Współczesnej J. M. Jasnorzewska, Lodz
  - NeuroMed, Lublin
  - Med Polonia Sp z o.o., Poznan
  - Centrum Medyczne Mrukmed, Rzeszów
  - Centrum Medyczne Pratia, Skorzewo
  - Wojewodzki Szpital Zespolony im. L. Rydygiera w Toruniu, Oddzial Chemioterapii Nowotworow, Torun
- Taiwan (7):
  - Taipei Veterans General Hospital, Taipei, Beitou District
  - Chang-Gung Memorial Hospital - Linko, Taoyuan, Guishan District
  - Tri-Service General Hospital, Taipei, Neihu District
  - Chang-Gung Memorial Hospital, Kaohsiung City, Niaosong District
  - Taipei Tzu Chi Hospital, New Taipei City, Xindian Dist
  - Taipei Medical University Hospital, Taipei, Xinyi District
  - National Taiwan University Hospital, Taipei, Zhongzheng District
- Turkey (Türkiye) (2):
  - Liv Hospital Ankara, Medikal Onkoloji Bilim Dalı, Ankara
  - İstinye Üniversitesi Hastanesi Liv Hospital Bahçeşehir, Istanbul

IPD SHARING:
Plan to Share IPD: No